CLINICAL TRIAL: NCT04205656
Title: Prospective Evaluation of Platelet-Rich Plasma and Bone Marrow Concentrate Treatment to Accelerate Healing After Anterior Cruciate Ligament Reconstruction
Brief Title: Prospective Evaluation of PRP and BMC Treatment to Accelerate Healing After ACL Reconstruction
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Steadman Philippon Research Institute (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Office of Naval Research (ONR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-13
Record Dates: First submitted 2019-12-04; First posted 2019-12-19 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Osteoarthritis, Knee
Keywords: bone marrow concentrate (BMC); stem cell; platelet-rich plasma (PRP); anterior cruciate ligament reconstruction (ACLR)
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Leukocyte-Poor Platelet Rich Plasma (LP-PRP) (Experimental): Participants will have a knee injected with Platelet-Rich Plasma (PRP) obtained from a venous whole blood draw from the vein.
  Interventions: Biological: Leukocyte-Poor Platelet Rich Plasma (LP-PRP)
- Bone Marrow Concentrate (BMC) (Experimental): Participants will have a knee injected with BMC stem cells harvested from the iliac crest
  Interventions: Biological: Bone Marrow Concentrate (BMC)
- Control (Placebo Comparator): Patients randomized in the placebo arm will undergo their standard of care treatment and will not receive LP-PRP or BMC.
  Interventions: Other: Control group (Placebo)

INTERVENTIONS:
Biological: Leukocyte-Poor Platelet Rich Plasma (LP-PRP) — Participants will have a knee injected with Platelet-Rich Plasma (PRP) obtained from a venous whole blood draw from the vein.
  Arms: Leukocyte-Poor Platelet Rich Plasma (LP-PRP)
Biological: Bone Marrow Concentrate (BMC) — Participants will have a knee injected with BMC stem cells harvested from the iliac crest
  Arms: Bone Marrow Concentrate (BMC)
Other: Control group (Placebo) — Participants will undergo ACLR surgery with no injection into their knee.
  Arms: Control

SUMMARY:
This is a prospective, randomized, placebo-controlled trial to evaluate potential beneficial effects of leukocyte-poor platelet rich plasma and bone marrow concentrate on the healing and health of critical joint tissues in the knee following anterior cruciate ligament (ACL) reconstruction. Bone marrow contains stem cells which can change into cells of various different tissue types, while platelet rich plasma contains growth factors. This trial will compare the two procedures against placebo.

DETAILED DESCRIPTION:
This is a prospective, randomized, placebo-controlled trial. Patients will be randomized into three groups: Concentrated Bone Marrow Concentrate (BMC), Platelet-Rich Plasma (PRP) or Placebo. BMC subjects will have bone marrow aspirated from the subjects iliac crests and the cellular rich portion will be concentrated and subsequently injected into the subjects' symptomatic knee during ACL reconstruction surgery. PRP subjects will have a venous blood draw and the resulting PRP will be injected into the symptomatic knee during ACL reconstruction surgery. Follow-up visits in person will take place at 2 weeks, 6 months and 12 months after the ACL reconstruction surgery.

The purpose of this study is to evaluate potential beneficial effects of leukocyte-poor platelet-rich plasma (LP-PRP) and bone marrow concentrate (BMC) on the healing and health of all critical joint tissues (grafts/ligaments, meniscus and cartilage) in the knee following anterior cruciate ligament reconstruction (ACLR). Key aspects of this proposal include our well-developed methodologies to quantify and correlate cytokines, chemokines, growth factors in PRP and progenitor cells in BMC, clinical outcomes and imaging following ACLR. The overarching goal of this randomized control trial is to establish a biological signature of PRP and BMC that will be indicative for optimal recovery after ACLR. The long-term goal of our research is to better understand the efficacy of orthobiologic approaches to improve clinical outcomes, enhance graft healing and mitigate post-traumatic osteoarthritis (PTOA) in a cohort of patients that have undergone ACLR.

ELIGIBILITY:
Inclusion Criteria: Subjects will be included if all the following criteria are met:

1. Age 16-50 years at the time of Anterior Cruciate Ligament Reconstruction (ACLR) surgery;
2. Acute ACL injury within 6 months of scheduled ACLR surgery;
3. Scheduled for unilateral, primary ACLR with a BTB (bone-patellar tendon-bone) autograft;
4. The following concomitant injuries are allowed:

   1. Meniscal injuries of all types, grades and regardless of surgical treatment;
   2. Articular chondral injury that can be addressed with debridement or chondroplasty;
   3. Tibial impaction fractures;
   4. Non-operative sprains/injuries of MCL or LCL;
5. Willing and able to comply with all required post-operative visits, biomotion and imaging tests, the self-completion of questionnaires and other trial procedures.

Exclusion Criteria: Subjects will be excluded if any of the following criteria are met:

1. Inability to provide informed consent;
2. Women who are pregnant;
3. Previous surgery for either knee except in cases of prior diagnostic arthroscopy and/or minimal debridement;
4. Significant osteoarthritis (OA) of the knee (e.g. grade 4 with cystic changes and/or significant osteophytes);
5. Concomitant cartilage restoration procedure in the operative knee;
6. Biologic treatment (e.g. PRP, BMC, prolotherapy, etc.) in the operative knee within 6 months of ACLR surgery;
7. Steroid injections in the operative knee within 3 months of ACLR surgery;
8. Open growth plates (determined by the treating physician based on standard-of-care preoperative knee radiographs);
9. History of deep vein thrombosis (DVT) or pulmonary embolism (PE) that requires additional anticoagulation beyond usual post-operative standard of care;
10. Current or known history of significant active autoimmune disease (i.e. rheumatoid arthritis and SLE);
11. Incompatible MRI hardware/devices and/or inability to safely undergo MRI per the MRI safety screening questionnaire;
12. Known balance or vestibular disorders, if in the opinion of the Principal Investigator or delegated clinician may affect ability to safely comply with study procedures;
13. History of significant radiation exposure, e.g. due to radiation therapy or occupational exposure;
14. Active malignancy of any type or history of a malignancy within 2 years of informed consent (with the exception of subjects with a history of treated basal or squamous cell carcinoma);
15. Concurrent or previous participation in another clinical trial within 30 days prior to informed consent;

    1. Concurrent enrollment in DOD Project 4, Vail Health Hospital IRB # 2018-20, is allowed while subjects on this study are in the 18-month follow-up period;
    2. Concurrent enrollment in non-interventional registry studies or blood-banking/biomarker studies is allowed;
16. History of substance abuse (drug or alcohol) that may interfere with the subject's ability to cooperate and comply with the trial procedures;
17. Severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the Principal Investigator or delegated clinician, would make the subject inappropriate for entry into this trial.

    Subjects will be withdrawn from the study (Screen Failures) after providing informed consent and/or at the time of ACLR surgery if they meet any of the following criteria:
18. Concurrent reconstruction of any knee ligaments other than the ACL;
19. ACLR which requires the following concomitant treatments: bone plating, metal implants (with the exception of titanium interference screws) or microfracture;
20. Inability to collect sufficient research samples (e.g. less than the minimum required amount of BMA is harvested, or clotting occurs).

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 18 months
  Occurrence of adverse events

SECONDARY OUTCOMES:
Patient reported outcome questionnaire | screening, baseline, two weeks post-surgery, then every week for 8 weeks post-surgery; 3, 6 12 and 18 months post-surgery
  SF-12 Short Form General Health Survey Patient Satisfaction
Measure signature cellular profile of BMC | Day of Surgery
  Flow cytometer to analyze BMC cell concentrations
Measure plasma levels of pro-inflammatory factors in BMC | Day of Surgery
  Multiplex analysis of pro-inflammatory cytokines and chemokines using Luminex 200®
Measure plasma levels of pro-inflammatory factors in LP-PRP | Day of Surgery
  Multiplex analysis of pro-inflammatory cytokines and chemokines using Luminex 200®
Quantitative Magnetic Resonance Imaging (MRI) | screening, baseline; 6 and 12 months post-surgery
  Images acquired on a 3T Siemens Magnetom Skyra-fit scanner
DSX: three dimensional (3D) to measure motion of the knee using dynamix x-ray software | 6 and 12 months post-surgery
  Up to three brief X-ray exposures (6 scouts x 3 frames and 2 statics x 5 frames and 24 exposures x 100 frames will be acquired)
Computerized tomography (CT): 3D geometry of bony anatomy using a series of x-rays | 6 months post-surgery
  single, bilateral knee CT scan using Toshiba Aquilon Premium 160 CT scanner
Patient Reported Outcome questionnaire | screening, baseline, two weeks post-surgery, then every week for 8 weeks post-surgery; 3, 6 12 and 18 months post-surgery
  IKDC - International Knee Documentation Committee Score
Patient Reported Outcome questionnaire | screening, baseline, two weeks post-surgery, then every week for 8 weeks post-surgery; 3, 6 12 and 18 months post-surgery
  WOMAC - Western Ontario & McMaster Universities Osteoarthritis Index
Patient Reported Outcome questionnaire | screening, baseline, two weeks post-surgery, then every week for 8 weeks post-surgery; 3, 6 12 and 18 months post-surgery
  Lysholm Score
Patient Reported Outcome questionnaire | screening, baseline, two weeks post-surgery, then every week for 8 weeks post-surgery; 3, 6 12 and 18 months post-surgery
  Tegner Activity Scale
Patient Reported Outcome questionnaire | screening, baseline, two weeks post-surgery, then every week for 8 weeks post-surgery; 3, 6 12 and 18 months post-surgery
  NRS (NUMERICAL RATING SCALE) for Pain
Motion Assessment | screening, baseline; 6 months post-surgery
  3D video motion capture

CONTACTS AND LOCATIONS:
Overall Officials: Peter Millett, MD, Principal Investigator — The Steadman Clinic
Locations (1):
- 181 West Meadow Drive, Suite 1000, Vail, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided